CLINICAL TRIAL: NCT00616616
Title: Single Incision Laparoscopy
Acronym: SIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071271
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Appendicitis; Cholelithiasis; Malignant Hypertension
Keywords: appendectomy; cholecystectomy; gastric banding; adrenalectomy; Gastric lap-band placement
MeSH Terms: conditions — Appendicitis; Cholelithiasis; Hypertension, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): all subjects
  Interventions: Procedure: single incision laparoscopic surgery

INTERVENTIONS:
Procedure: single incision laparoscopic surgery — Surgery will be performed with ine laparoscopic incision

SUMMARY:
Laparoscopic surgery being performed with only one small incision via the umbilicus (belly button).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. Patient has consented for a laparoscopic operation (independent of study participation)
3. Attending surgeon decides operation can be completed via a single incision laparoscopic approach

Exclusion Criteria:

1. Patients with BMI greater than 40
2. Minors and cognitively impaired individuals
3. Patients who are ASA class IV - Illness that is a constant threat to life
4. Patients with ascites or Child's class C of liver failure
5. Patients with known common bile duct stones
6. Patients with coagulopathy, abnormal coagulation studies, or who take heparin, coumadin, Plavix (clopidogrel), aspirin, or other medication for the purpose of anti-coagulation and cannot be removed from the medication prior to the operation.
7. Patients who present with incarcerated (irreducible) or strangulated hernias
8. Patients with preoperative hematocrits less than 25.
9. Preoperative hematocrit less than 25.
10. Patients who have evidence of hemodynamic instability including systolic blood pressure greater than 200 or less than 80.
11. Heart rate greater than 130 or less than 50. Respiratory rate greater than 35 or less than 6. Patients who are on continuous pressor drip for blood pressure support.
12. Patients who present for emergency adrenalectomy.
13. Patients with CT scan evidence of an abdominal abscess.
14. Patients who present 48 hours after the onset of abdominal pain (appendectomy patients)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and efficacy of single incision laparoscopy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States